CLINICAL TRIAL: NCT03738020
Title: A Randomized, Multi Center, Single-blind, Active-controlled, Matched Pairs Design Clinical Study to Evaluate the Correction of Wrinkles and Folds and Safety of HA IDF Versus Restylane in Nasolabial Fold Intradermal Injection
Brief Title: Clinical Study to Evaluate the Correction of Wrinkles and Folds and Safety of YVOIRE Classic Versus Restylane in Nasolabial Fold Intradermal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-HACL008
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Temporary Correction of Wrinkles

STUDY DESIGN:
Intervention Model Description: IND approved from KFDA
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA IDF (Experimental)
  Interventions: Device: HA IDF (YVOIRE classic)
- Restylane (Active Comparator)
  Interventions: Device: Restylane

INTERVENTIONS:
Device: HA IDF (YVOIRE classic) — Treatment with HA IDF
  Arms: HA IDF
Device: Restylane — Treatment with Restylane
  Arms: Restylane

SUMMARY:
This study was purposed to evaluate the non-inferiority of HA IDF, a hyaluronic acid product, in terms of correction of wrinkles and safety in nasolabial fold intradermal injection, compared to Restylane, the control preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Women in 30~55 years.
2. Those whose wrinkle scores in the treatment site (nasolabial fold) at the screening visit were Stage 3 or 4 in the 5-stage Wrinkle Severity Rating Scale (WSRS) symmetrically and who were informed on this study in detail, understood it completely, decided to participate in the study own their own and signed on the informed consent.

Exclusion Criteria:

1. Those with a skin disease in the face (skin infection, eczema, psoriasis, rosacea, herpes etc.) or those with a history of severe allergy.
2. Patients with a disorder in autoimmune system
3. Those with hepatic dysfunction or abnormality in coagulation, or those administering an anticoagulant (aspirin, warfarin etc.) concomitantly
4. Those who had used a local topical preparation (steroid, retinoid) within 4 weeks prior to the study.
5. Those who had underwent a chemical peeling, laser procedure (including IPL) or insertion of other bioadaptive material within 3 months prior to the study (however, those who had been treated with HA filler could participate in the study if the date of treatment was known and the investigator judged that the filler effect had disappeared).
6. Patients with a malignant tumor
7. Women in pregnancy or lactation
8. Hepatitis carriers or VDRL/HIV positive patients
9. Those with a hypersensitivity to the investigational medical device of this study
10. Other persons including those considered as difficult to perform this study by the principal investigator

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: spilt-face design
Groups:
- Subjects: Subjects who enrolled in this study
Period: Overall Study
Arm/Group | Subjects
Started | 58
Completed | 57
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: spilt-face design
Groups:
- HA IDF and Restylane: Subjects who were included in efficacy evaluation
Arm/Group | HA IDF and Restylane
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.40 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 58

OUTCOME MEASURES:

1. Primary Outcome: Average of Wrinkle Severity Rating Scale (WSRS) Score Evaluated by the Evaluating Investigator at Week 26 (Visit 7) After the Final Treatment With the Investigational Medical Device
Description: Wrinkle Severity Rating Scale (WSRS)
  1. Absent: no visible fold; continuous line
  2. Mild: Shallow but visible fold with slight indentation; minor facial feature
  3. Moderate: moderately deep fold; clear facial feature visible at normal appearance but not when stretched. Excellent correction expected.
  4. Severe: very long and deep; prominent facial feature; less than 2mm visible fold when stretched
  5. Extreme: extremely deep and long folds; 2-4mm visible v-shaped fold when stretched; detrimental to appearance; unlikely to have satisfactory correction with injectable implant alone
Time Frame: Week 26 (Visit 7)
Population: Spilt-face design
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HA IDF | Restylane
Number analyzed (Participants) | 58 | 58
score on a scale | 2.56 (0.68) | 2.56 (0.66)

ADVERSE EVENTS:
Groups:
- HA IDF; Restylane; Systemic: Subject who were injected with investigational medical device at least once
Arm/Group | HA IDF | Restylane | Systemic
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 3/58 | 3/58 | 5/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HA IDF (N=58) | Restylane (N=58) | Systemic (N=58)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 5
Application site erythema (General disorders) | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other